CLINICAL TRIAL: NCT01690897
Title: Randomized Comparison of Mindfulness Versus Group Support for Treatment of Low Sexual Desire in Women
Acronym: DESIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Professor, UBC Department of Gynaecology, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12-01659
Record Dates: First submitted 2012-08-22; First posted 2012-09-24 (Estimated); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Low Female Sexual Desire
Keywords: Female sexual desire; Psychoeducational intervention; Mindfulness
MeSH Terms: interventions — Educational Status

ARMS (2):
- MBCT group (Experimental): Women randomized into the MBCT group will undergo pre-treatment testing (questionnaires, saliva sample collection, and physiological assessment) within 2.5 months of beginning the mindfulness-based treatment.
  Interventions: Behavioral: Mindfulness-based treatment
- Support group (Active Comparator): Women randomized into the support group will undergo pre-treatment testing (questionnaires, saliva sample collection, and physiological assessment) within 2.5 months of beginning the sex therapy, education, and support treatment.
  Interventions: Behavioral: Sex therapy, education, and support treatment

INTERVENTIONS:
Behavioral: Mindfulness-based treatment — The mindfulness-based treatment for the MBCT group treatment consists of eight 2-hour long weekly sessions, based on a variety of empirically supported techniques, and integrates elements of education, mindfulness skills, and sex therapy. In addition, participants are also given handouts and asked to complete approximately 10-60 minutes/day of at-home practice/skills, which may include reading material, mindfulness exercises, and behavioural exercises between sessions.
  Arms: MBCT group
Behavioral: Sex therapy, education, and support treatment — The sex therapy, education, and support group will consist of all of the same techniques and materials in the MBCT group except for the mindfulness components in group sessions and at-home practices.
  Arms: Support group

SUMMARY:
The purpose of this study is to determine whether an 8-session mindfulness-based intervention (MBCT group) is effective for women with low sexual interest/desire in reducing sexual distress, improving their sexual response, and increasing their mindful skills, compared to a support group.

DETAILED DESCRIPTION:
HYPOTHESES:

1. Compared to baseline, the MBCT group will have significant post-treatment improvements in self-report measures of: (a) sexual distress; (b) sexual desire, subjective sexual arousal, perception of genital arousal, and sexual pleasure; (c) relationship satisfaction; (d) depressive symptoms and rumination; (e) perceived stress, general anxiety, anxiety sensitivity, and sexuality-related situational anxiety (as self-reported at the sexual arousal assessment); and (f) mindfulness, self-compassion, non-attachment, and interoceptive awareness.
2. Compared to baseline, the MBCT group will have significant post-treatment improvements in laboratory physiological measures of: (a) genital sexual response as measured by a vaginal photoplethysmograph, (b) interoceptive awareness, as measured by a heart rate perception task, and (c) cortisol:DHEA ratio as measured by hormonal assays of saliva samples.
3. We hypothesize that the changes in the endpoints listed in #1 or #2 will be significantly greater in the MBCT group than in the support group.
4. We hypothesize that participation in the MBCT group will significantly increase concordance between genital and subjective sexual arousal.
5. Mindfulness, self-compassion, and interoceptive awareness will significantly mediate improvements in sexual distress and desire in the MBCT group at all post-treatment assessment points.
6. Expectations of change with treatment will not significantly moderate improvements in sexual distress and desire in the MBCT group.
7. Participants' impressions of change will be significantly greater in the MBCT group compared to the support group at all post-treatment assessment points.
8. We hypothesize that participants will experience fewer breaks in the sexual response cycle throughout the course of the eight-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* must be experiencing distressing sexual interest/desire and/or sexual arousal concerns
* must between the ages of 19 - 65
* must be fluent in English

Exclusion Criteria:

* not experiencing distressing sexual interest/desire and/or sexual arousal concerns
* not between the ages of 19-65
* unable to read, write, speak and understand English

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Department of Gynaecology, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Brotto LA, Basson R, Grabovac A, Chivers ML, Zdaniuk B, Bodnar TS, Weinberg J. Impact of mindfulness versus supportive sex education on stress in women with sexual interest/arousal disorder. J Behav Med. 2024 Aug;47(4):721-733. doi: 10.1007/s10865-024-00491-5. Epub 2024 Apr 26. PMID 38668816
- [Derived] Brotto LA, Zdaniuk B, Chivers ML, Jabs F, Grabovac A, Lalumiere ML, Weinberg J, Schonert-Reichl KA, Basson R. A randomized trial comparing group mindfulness-based cognitive therapy with group supportive sex education and therapy for the treatment of female sexual interest/arousal disorder. J Consult Clin Psychol. 2021 Jul;89(7):626-639. doi: 10.1037/ccp0000661. PMID 34383535

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MBCT Group | Support Group
Started | 70 | 78
Completed | 55 | 59
Not Completed | 15 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBCT Group | Support Group | Total
Number analyzed (Participants) | 70 | 78 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (13.2) | 37.9 (12.2) | 38.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 78 | 148
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 67 | 71 | 138
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 70 | 78 | 148
Sexual Interest/Desire Inventory (SIDI) [Mean (Standard Deviation); unit: units on a scale] — Sexual Interest and Desire Inventory (SIDI) is a 14-item questionnaire that assesses sexual desire in women which includes one non-scored item assessing intercourse frequency. Possible total scores range from 0 - 51, with higher scores indicating higher levels of sexual functioning. Scoring Instruction: Sum total of all items [Scores Range: 1 - 51]. Outcomes shown are mean of group scores. Population: Numbers assessed at baseline differed due to participants lost before treatment started or did not complete.
  units on a scale
    number analyzed (Participants) | 64 | 69 | 133
    (all) | 16.99 (8.16) | 15.41 (6.66) | 16.17 (7.43)
Female Sexual Distress Scale-Revised (FSDS-R) [Mean (Standard Deviation); unit: units on a scale] — The Female Sexual Distress Scale (FSDS) is a 12-item self-report questionnaire assessing for sexuality related personal distress. Scores on the scale range from 0 - 48, where higher scores represent higher levels of distress. The FSDS has been shown to have good discriminant validity in differentiating between sexually dysfunctional and sexually functional women, with 88% correct classification rate. Scores on the scale range from 0 - 48, where higher scores represent higher levels of distress. Population: Numbers assessed at baseline differed due to participants lost before treatment started or did not complete.
  units on a scale
    number analyzed (Participants) | 64 | 69 | 133
    (all) | 32.97 (11.27) | 32.22 (7.99) | 32.58 (9.68)
Relationship Assessment Scale (RAS) [Mean (Standard Deviation); unit: units on a scale] — The Relationship Assessment Scale (RAS) was designed to assess to measure an individual's satisfaction with their relationship. Relationship satisfaction is one of the key areas of relationship assessment. The RAS is a brief measure of global relationship satisfaction. It consists of seven items, each rated on a five-point likert scale. Scoring: Add up the 7 item scores and divide by 7 to get a mean score. Minimum score 1, maxiumum score 5. Higher score means higher satisfaction. Population: Numbers assessed at baseline differed due to participants lost before treatment started or did not complete.
  units on a scale
    number analyzed (Participants) | 64 | 69 | 133
    (all) | 3.87 (0.80) | 4.14 (0.74) | 4.01 (0.77)
Rumination-Reflection Questionnaire (RRQ) [Mean (Standard Deviation); unit: units on a scale] — Rumination was measured with the Rumination-Reflection Questionnaire - Adapted Rumination Subscale (adapted from Trapnell & Campbell, 1999 to inquire about sexuality-related rumination). Likert scale 1 - 5 with higher score indicating higher rumination. Population: Numbers assessed at baseline differed due to participants lost before treatment started or did not complete.
  units on a scale
    number analyzed (Participants) | 64 | 69 | 133
    (all) | 3.08 (.96) | 3.00 (.79) | 3.04 (.87)

OUTCOME MEASURES:

1. Primary Outcome: Female Sexual Distress Scale-Revised (FSDS-R)
Description: Sexual distress will be measured with the revised version of the Female Sexual Distress Scale-R (Derogatis et al., 2008). Scores on the scale range from 0 - 48, where higher scores represent higher levels of distress.
Time Frame: 2-4 weeks post treatment (10-12 weeks after start of treatment), 6 months post (approx 8 months after start), and 12 months post (approx 14 months after start of treatment). Assessments completed past 1 year were due to personal delays by co-investigator.
Population: Numbers adjusted due to participants lost before treatment, did not complete, scheduling difficulties, or removed from study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
units on a scale
  Post-treatment: number analyzed (Participants) | 61 | 68
  Post-treatment | 22.88 (10.73) | 25.68 (10.24)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 23.02 (11.54) | 23.87 (11.83)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 18.92 (9.63) | 21.60 (11.95)

2. Primary Outcome: Sexual Interest and Desire Inventory (SIDI)
Description: The Sexual Interest and Desire Inventory (SIDI; Clayton et al. 2006) will be used to measure sexual desire. Possible total scores range from 0 - 51, with higher scores indicating higher levels of sexual functioning.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
units on a scale
  Post treatment: number analyzed (Participants) | 61 | 68
  Post treatment | 27.91 (9.81) | 23.62 (9.91)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 28.08 (10.44) | 25.57 (10.77)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 29.85 (9.78) | 26.76 (11.51)

3. Primary Outcome: Rumination
Description: Rumination was measured with the Rumination-Reflection Questionnaire - Adapted Rumination Subscale (adapted from Trapnell & Campbell, 1999 to inquire about sexuality-related rumination). Likert scale 1 - 5 with higher score indicating higher rumination.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
units on a scale
  Post-treatment: number analyzed (Participants) | 61 | 68
  Post-treatment | 2.60 (.72) | 2.71 (.92)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 2.32 (.72) | 2.81 (1.01)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 2.23 (.72) | 2.47 (.99)

4. Primary Outcome: Relationship Assessment Scale (RAS)
Description: Relationship satisfaction will be measured with the Relationship Assessment Scale (Hendrick, 1988). Scoring: Add each item score and divide by 7 to get a mean score. Higher score relates to higher satisfaction. Minimum mean score 1, maximum score 5.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
units on a scale
  Post treatment: number analyzed (Participants) | 61 | 68
  Post treatment | 4.27 (0.71) | 4.03 (0.89)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 3.87 (.80) | 4.14 (.74)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 4.16 (.75) | 4.24 (.85)

5. Secondary Outcome: Subjective Sexual Arousal
Description: Subjects will indicate their levels of subjective arousal while undergoing arousal testing. A device manufactured for the UBC Sexual Health Lab called the "arousometer"- a computer mouse mounted on a metal track divided into 10 equally spaced intervals corresponding to "sexually turned off" (-2) to "the most sexually aroused you have ever been or could imagine being" (7). This device allows continuous self-report measurement of subjective sexual arousal while viewing the erotic films.
Time Frame: Up to 2 mos pre-treatment, 2-4 weeks post treatment (10-12 weeks after treatment start), 6 months post (approx 8 months after start), and 12 months post (approx 14 months after start). Assessments completed past 1 year were due to personal delays by Co-I
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
score on a scale
  Pre Treatment: number analyzed (Participants) | 64 | 69
  Pre Treatment | 2.96 (1.53) | 3.21 (1.37)
  Post Treatment: number analyzed (Participants) | 61 | 68
  Post Treatment | 3.93 (1.48) | 3.74 (1.4)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 3.8 (1.53) | 3.77 (1.53)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 3.78 (1.46) | 3.73 (1.59)

6. Secondary Outcome: Interoceptive Awareness
Description: Interoceptive awareness will be measured using the Multidimensional Assessment of Interoceptive Awareness (MAIA; Mehling et al., 2012) questionnaire. Possible range of scores 0 - 5. Higher score means higher awareness.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
score on a scale
  Pre Treatment: number analyzed (Participants) | 64 | 69
  Pre Treatment | 2.60 (.72) | 2.74 (.60)
  Post Treatment: number analyzed (Participants) | 61 | 68
  Post Treatment | 3.15 (.57) | 2.9 (.58)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 3.08 (.63) | 2.89 (.66)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 3.19 (.63) | 2.96 (.62)

7. Secondary Outcome: Physiological Sexual Arousal
Description: Physiological sexual arousal will be measured with a Vaginal Photoplethysmograph (VPP) during exposure to erotic films. The VPP measures vaginal pulse amplitude (VPA) which has been found to be a sensitive and specific measure of genital arousal (Laan & Everaerd, 1995). There is no threashold on the millivolts (MV) reading.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
millivolts (mV)
  Pre Treatment: number analyzed (Participants) | 64 | 69
  Pre Treatment | .120 (.093) | .125 (.091)
  Post Treatment: number analyzed (Participants) | 61 | 68
  Post Treatment | .124 (.099) | .135 (.100)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | .102 (.070) | .133 (.089)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | .119 (.095) | .151 (.100)

8. Secondary Outcome: Stress Hormone Cortisol Slope
Description: The diurnal cortisol slope is the difference in cortisol levels from morning to evening (PM minus AM). To assay salivary cortisol concentrations, samples were vortexed and centrifuged at 1,400 g for 10 minutes at 18°C. Salivary cortisol was measured using the commercially available High Sensitivity Salivary Cortisol Enzyme Immunoassay Kit (Salimetrics Assays, 1-3002, State College, PA) according to the standard protocol. The minimum amount of saliva required by this assay is 25 μl, and intra- and inter-assay coefficients of variation were 4.6% and 6.0%, respectively.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms per decilitre (ug/dl)
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
micrograms per decilitre (ug/dl)
  Pre Treatment: number analyzed (Participants) | 64 | 69
  Pre Treatment | .298 (.062) | .296 (.063)
  Post Treatment | .285 (.103) | .283 (.071)
  6 Months | .325 (.139) | .310 (.087)
  12 Months | .309 (.094) | .287 (.089)

9. Other Pre Specified Outcome: Depression
Description: Depression is measured with the Hamilton Depression Scale - Short Form (McIntyre et al., 2005). Seven questions on a scale of 0 - 4 with higher score meaning higher depression. Totals are summed with a possible range of scores from 0 - 28.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
score on a scale
  Pre Treatment: number analyzed (Participants) | 64 | 69
  Pre Treatment | 4.44 (3.47) | 4.70 (3.62)
  Post Treatment: number analyzed (Participants) | 61 | 68
  Post Treatment | 2.99 (2.49) | 3.95 (3.79)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 2.85 (3.18) | 3.47 (3.60)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 2.56 (2.91) | 3.54 (3.13)

10. Other Pre Specified Outcome: Mindfulness
Description: Mindfulness will be measured with the Five Factor Mindfulness questionnaire (Baer, Smith, Hopkins, Krietemeyer & Tony, 2006). Questions are answered on a 5-point Likert scale ranging from 1 to 5. Possible range of scores 39 to 195 with higher score meaning higher mindfulness.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
score on a scale
  Pre Treatment: number analyzed (Participants) | 64 | 69
  Pre Treatment | 123.76 (18.02) | 126.02 (17.95)
  Post Treatment: number analyzed (Participants) | 61 | 68
  Post Treatment | 134.47 (17.49) | 126.19 (17.67)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 131.92 (17.79) | 127.66 (19.16)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 138.06 (18.27) | 130.89 (19.35)

11. Other Pre Specified Outcome: Perceived Stress
Description: Perceived stress will be measured with the Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983). Questions are likert scale from 0 - 4. Possible range of scores 0 - 40 with higher score indicating higher stress.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBCT Group | Support Group
Number analyzed (Participants) | 70 | 78
score on a scale
  Pre Treatment: number analyzed (Participants) | 64 | 69
  Pre Treatment | 16.34 (6.56) | 17.66 (6.07)
  Post Treatment: number analyzed (Participants) | 61 | 68
  Post Treatment | 14.1 (6.25) | 16.5 (7.6)
  6 Months: number analyzed (Participants) | 58 | 63
  6 Months | 15.13 (6.55) | 15.46 (7.39)
  12 Months: number analyzed (Participants) | 55 | 59
  12 Months | 12.99 (6.14) | 16.51 (7.46)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at 2-4 weeks post treatment (10-12 weeks from start of treatment), 6 months post treatment (8 months from start of treatment), and at 12 months post treatment (14 months from start of treatment).
Description: Participants were asked if they had experienced any struggles or concerns during the post treatment assessments.
Arm/Group | MBCT Group | Support Group
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/78
Other Adverse Events (participants affected / at risk) | 0/70 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT01690897/Prot_SAP_000.pdf